CLINICAL TRIAL: NCT03017092
Title: Tobacco Pilot Study for Low Income Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-1442; 1R35CA197573-01 (NIH); A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison)
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2017-05

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tablet-guided (Experimental): Study participants will be administered a brief tobacco intervention by a Salvation Army staff person who is guided by a tablet computer
  Interventions: Behavioral: Tablet-guided tobacco intervention

INTERVENTIONS:
Behavioral: Tablet-guided tobacco intervention — This intervention, as guided by a tablet computer, is a brief (20 minute) counseling intervention designed to increase motivation to quit smoking and to increase knowledge of methods of quitting.

SUMMARY:
Pilot study to test feasibility of delivering a motivational smoking cessation intervention to low income smokers via a computer tablet.

DETAILED DESCRIPTION:
Twenty Salvation Army clients will be recruited to pilot test a motivational smoking cessation counseling intervention that is delivered via a tablet computer. Study participants will be given brief instructions on how to use the tablet. They will then complete a brief survey on the tablet. This will be followed by the researcher using the tablet to provide the motivational intervention. Finally, study participants will be interviewed to establish this perceptions of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* current smoker (≥ 10 cigarettes/week for the past six months who are not currently trying to quit)
* age ≥ 18 years
* English speaking/writing

Exclusion Criteria:

* not receiving services for the Salvation Army

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Ease of use of tablet-guided tobacco intervention assessed by interview and summarized across study participants | Immediately after exposure to intervention
  At the end of the intervention, each study participant will be interviewed regarding how easy the tablet computer was to use. This qualitative information will by summarized across all study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States